### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title

: Reporting and Analysis Plan for A Phase I, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Dolutegravir + Rilpivirine (JULUCA<sup>TM</sup>) 50 mg/25 mg tablets in healthy volunteers of Japanese descent

Compound Number : GSK3365791

Effective Date : 13-JUNE-2019

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 212312 [2018N392977\_00].
- This RAP will be provided to the study team members to convey the content of the 212312 Statistical Analysis Complete (SAC) deliverable.

### **RAP Author(s):**

| Approver | Date |
|----------------------------------------|-------------|
| PPD | 11-JUN-2019 |
| Principal Statistician (Biostatistics) | 11-JUN-2019 |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals (Method: E-mail):**

| Approver | Date | Approval Method |
|---|---|---|
| Senior Director, Clinical Pharmacology | 12-JUN-2019 | E-mail |
| Clinical Development Director, Global Medical | 12-JUN-2019 | E-mail |
| Medical Director, Global Clinical Safety and Pharmacovigilance | 12-JUN-2019 | E-mail |
| Principal Clinical Data Manager, Infectious Disease | 11-JUN-2019 | E-mail |
| Clinical Development, Infectious Disease | 12-JUN-2019 | E-mail |
| Programmer, Clinical Programming | 11-JUN-2019 | E-mail |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF eSignature):

| Approver | Date | Approval Method |
|---|---|---|
| * Statistics Director, Clinical Statistics | 13-JUN-2019 | e-signature |
| PPD ** Programming Manager, Clinical Programming | 13-JUN-2019 | e-signature |

<sup>\*</sup>Delegated to PPD , Statistics Leader by PPD , Statistics Director

<sup>\*\*</sup>Delegated to PPD , Programming Director

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 5 |
| 2. | CLIMAN | MARY OF KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| 3. | PLAN | NED ANALYSES | 6 |
| | 3.1. | Final Analyses | 6 |
| 4. | ANAL | YSIS POPULATIONS | 6 |
| | 4.1. | Protocol Deviations | 7 |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING /ENTIONS | Q |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 0 | 5.2.1. Derivations and Handling of Missing Baseline Data | |
| | 5.3. | Other Considerations for Data Analyses and Data Handling Conventions | |
| | | CONVENTIONS | |
| 6. | STUD | Y POPULATION ANALYSES | 11 |
| | 6.1. | Overview of Planned Study Population Analyses | 11 |
| 7. | SAFE | TY ANALYSES | 12 |
| | 7.1. | Adverse Events Analyses | |
| | 7.2. | Clinical Laboratory Analyses | 12 |
| | 7.3. | Other Safety Analyses | 13 |
| 8. | PHAR | RMACOKINETIC ANALYSES | 14 |
| | 8.1. | Primary Pharmacokinetic Analyses | 14 |
| | | 8.1.1. Overview of Planned Pharmacokinetic Analyses | 14 |
| | | 8.1.2. Endpoint / Variables | 14 |
| | | 8.1.2.1. Drug Concentration Measures | 14 |
| | | 8.1.2.2. Derived Pharmacokinetic Parameters | |
| | | 8.1.3. Population of Interest | 15 |
| | | 8.1.4. Statistical Analyses / Methods | 15 |
| 9. | REFE | RENCES | 17 |
| 10. | APPE | NDICES | 18 |
| | 10.1. | | |
| | | 10.1.1. Exclusions from PK Population | |
| | 10.2. | Appendix 2: Schedule of Activities | 19 |
| | | 10.2.1. Protocol Defined Schedule of Events | 19 |
| | 10.3. | Appendix 3: Study Phases | |
| | | 10.3.1. Study Phases | 21 |

| 10.3.2. | Study Phases for AE Data | 21 |
|---|---|---|
| Appendi | x 4: Data Display Standards & Handling Conventions | 22 |
| 10.4.1. | | |
| 10.4.2. | | |
| 10.4.3. | | |
| Appendi | | |
| 10.5.1. | | |
| 10.5.2. | Study Population | 24 |
| 10.5.3. | | |
| Appendi | <b>J</b> | |
| 10.6.1. | | |
| 10.6.2. | Handling of Missing Data | 26 |
| Appendi | | |
| 10.7.2. | | |
| 10.7.3. | Vital Signs | 28 |
| 10.8.1. | | |
| 10.8.2. | Trademarks | 30 |
| Appendi | x 9: List of Data Displays | 31 |
| 10.9.1. | • • | |
| 10.9.2. | | |
| 10.9.3. | | |
| 10.9.4. | | |
| 10.9.5. | | |
| 10.9.7. | <u> </u> | |
| 10.9.8. | Non-ICH Listings | |
| | Appendi<br>10.4.1.<br>10.4.2.<br>10.4.3.<br>Appendi<br>10.5.1.<br>10.5.2.<br>10.5.3.<br>Appendi<br>10.6.1.<br>10.6.2.<br>Appendi<br>10.7.3.<br>Appendi<br>10.8.1.<br>10.8.2.<br>Appendi<br>10.9.1.<br>10.9.2.<br>10.9.3.<br>10.9.4.<br>10.9.5.<br>10.9.6.<br>10.9.7. | 10.4.2. Reporting Standards 10.4.3. Reporting Standards for Pharmacokinetic. Appendix 5: Derived and Transformed Data 10.5.1. General |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 212312:

| Revision Chronology: | | |
|----------------------|-------------|----------|
| Original | 04-APR-2019 | Original |
| Document | | |
| Number | | |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol [(Dated: 04/APR/2019)].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the PK of DTG and<br>RPV following a single oral<br>dose of DTG/RPV 50 mg/25<br>mg FDC in healthy, adult<br>Japanese participants. | <ul> <li>Plasma DTG and RPV AUC<sub>(0-∞)</sub>, AUC<sub>(0-t)</sub>, C<sub>max</sub>, t<sub>lag</sub>, t<sub>max</sub>, t, t<sub>½</sub>, λz, %AUC<sub>ex</sub>, AUC<sub>(0-24)</sub>, AUC<sub>(0-72)</sub>, CL/F and Vz/F, C<sub>t</sub>, and C<sub>24</sub> following a single oral dose of DTG/RPV 50 mg/25 mg FDC in healthy adult Japanese participants.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the safety and tolerability of DTG/RPV FDC in healthy, adult Japanese participants. | Safety and tolerability parameters, adverse event (AE) /serious adverse events (SAE), observed and change from baseline clinical laboratory values, and vital sign assessments. |

# 2.3. Study Design

| Design<br>Features | • This is a single dose, open-label study in adult Japanese healthy participants to evaluate the PK, safety and tolerability of DTG/RPV 50 mg/25 mg FDC tablets. The study will consist of screening, treatment and follow-up phases. |
|---|---|
| Dosing | • Enrolled participants will receive the DTG/RPV 50 mg/25 mg FDC tablet as a single oral dose in a fed state. |
| Time & Events | Refer to Appendix 2: Schedule of Activities |
| Treatment<br>Assignment | • A maximum of 16 healthy adult Japanese subjects will be randomized such that a minimum of approximately 13 evaluable subjects complete the study with at least 3 participants of each gender enrolled. |
| Interim<br>Analysis | There will be no interim analysis. |

See study protocol for further details

# 2.4. Statistical Hypotheses / Statistical Analyses

This study is designed to characterize the pharmacokinetics of DTG and RPV following a single oral dose of DTG/RPV 50 mg/25 mg FDC in healthy, adult Japanese subjects. Also, this study will seek to assess the safety and tolerability of DTG/RPV 50 mg/25 mg FDC in healthy, adult Japanese participants.

No formal statistical hypothesis will be tested.

### 3. PLANNED ANALYSES

# 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who sign the ICF | <ul><li>Screen Failures</li><li>Protocol<br/>Deviations</li></ul> |
| Enrolled | All participants who have a Day 1 visit. | Study Populations |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Safety | All participants who enrolled in the study and received at least one dose of study drug. | <ul><li>Study Population</li><li>Safety</li></ul> |
| Pharmacokinetic (PK) | <ul> <li>All participants in the Safety population for whom a PK sample was obtained and had evaluable PK assay results.</li> <li>A subject with emesis occurring within 10 hours of the dose will not be considered evaluable.</li> </ul> | Data from subjects who vomit within 10 hours of study drug administration will be excluded from PK concentration summary and PK parameter summary but will be included in the listing and flagged. Excluded subjects will be flagged in footnotes for summary tables. |

Refer to Appendix 9 List of Data Displays which details the population used for each display.

# 4.1. Protocol Deviations

| Term | Definition |
|---|---|
| Study Deviation<br>Rules Document | The document describing study deviations (and associated coding/naming conventions) that may be identified during a study and the frequency of study deviation reviews. |
| Protocol Deviation (PD) | Any departure from study-specific requirements specified in a protocol. Subsets of protocol deviations are categorized as important or significant. |
| Important Protocol<br>Deviations | A subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or wellbeing. All-important deviations have a Violation Flag in CTMS and are associated with a Rule Number. |

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | |
|------------------------------|--------------|
| Data Displays for Reporting | |
| Description | Order in TLF |
| DTG/RPV 50mg/25mg FDC | 1 |

### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the last available assessment prior to time of the dose, unless noted otherwise. If there are multiple assessments collected on the same scheduled time, the average of these assessments will be used.

| Parameter | Study Asses | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | | | | |
| Labs | Х | X | | Day -1 |
| Vital Signs | Х | Х | X | Day 1 (Pre-Dose) |

# 5.2.1. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 5.2 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|-----------------------------------------------------------|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions |
| 10.2 | Appendix 2: Schedule of Activities |
| 10.3 | Appendix 3: Treatment States and Phases |
| 10.4 | Appendix 4: Data Display Standards & handling Conventions |
| 10.5 | Appendix 5: Derived and Transformed Data |
| 10.6 | Appendix 6: Reporting Standards for Missing data |
| 10.7 | Appendix 7: Values of Potential Clinical Importance |
| 10.8 | Appendix 8: Abbreviations & Trade Marks |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 1 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 9: List of Data Displays.

 Table 1
 Overview of Planned Study Population Analyses

| Display Type | Data Display's Generated | | |
|---|---|---|---|
| | Figure | Table | Listing |
| Randomisation | | | |
| Randomisation | | | Y |
| <b>Subject Disposition</b> | | | |
| Participant Disposition | | Y | |
| Reasons for Screen Failure | | Y | Y |
| Reasons for Withdrawals | | | Y |
| Important Protocol Deviations | | Y | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Subjects Excluded from Analysis Populations | | | Y |
| Medical history | | Y | |
| Demography | | | • |
| Demographics Characteristics | | Y | Y |
| Race and Racial Combinations | | Y | Y |
| Age Ranges | | Y | |
| <b>Concomitant Medications</b> | | | |
| Concomitant Medications | | | Y |

### 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

Table 2 Overview of Planned Safety Analyses

| Display Type | Absolute | | | Change from Baseline | | | е | |
|---|---|---|---|---|---|---|---|---|
| | Sun | nmary | Individual | | Summary | | Individual | |
| | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Exposure Data | | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| Relationship Between | | | | Υ | | | | |
| System Organ Class and | | | | | | | | |
| Verbatim Term | | | | | | | | |
| Subject Numbers for | | | | Υ | | | | |
| Individual AEs | | | | | | | | |
| All AEs | Υ | | | Υ | | | | |
| All Drug-Related AEs | Υ | | | Υ | | | | |
| Serious AEs | | | | Υ | | | | |
| Withdrawal AEs | | | | Υ | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual participant observed raw data.

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 9: List of Data Displays.

| Display Type | | Abs | solute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sur | nmary | Indiv | idual | Summary | | Individual | |
| | Т | F | F | L | T | F | F | L |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Υ | | | Υ [1] | Υ | | | |
| Hematology | Υ | | | Υ [1] | Υ | | | |
| Abnormal Chemistry | | | | Υ [1] | | | | |
| Abnormal Hematology | | | | Υ [1] | | | | |
| Urinalysis | Υ | | | Υ [1] | | | | |

| Electrocardiograms (ECC | Gs) | | |
|-------------------------|-----|--------------|---|
| ECG Findings | Υ | Υ [2] | |
| ECG Values | | Y [3] | |
| Vital Signs | | | |
| Vital Signs | Υ | <b>Y</b> [3] | Υ |
| Liver | | | |
| Liver Events [1] | | Υ | |

#### NOTES:

- 1. Displays contain only participants with DAIDS toxicities for HIV-infected patients
- 2. Displays contain only participants with abnormal findings
- 3. Displays contain only participants with values of potential clinical importance
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual participant observed raw data.

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9: List of Data Displays.

| Display Type | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sur | nmary | Indiv | idual | Sum | mary | Indiv | ridual |
| | Т | F | F | Ш | Т | F | F | L |
| Electrocardiograms (ECG | is) | | | | | | | |
| ECG Findings | Υ | | | Υ [2] | | | | |
| ECG Values | | | | Υ [3] | | | | |
| Vital Signs | | | | | | | | |
| Vital Signs | Υ | | | Y [3] | Υ | | | |
| Liver | | | | | | | | |
| Liver Events [1] | | | | Υ | | | | |

#### NOTES:

- 1. Displays contain only participants with DAIDS toxicities for HIV-infected patients
- 2. Displays contain only participants with abnormal findings
- 3. Displays contain only participants with values of potential clinical importance
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual participant observed raw data.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data. Individual = Represents TFL related to any displays of individual participant observed raw data.

# 8. PHARMACOKINETIC ANALYSES

# 8.1. Primary Pharmacokinetic Analyses

### 8.1.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK Population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 9: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untransformed | | | | Loge-1 | ransfor | med | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | Т | F | L | F | T | F | L |
| Plasma Drug Concentrations | <b>Y</b> [1] [2] | Υ | <b>Y</b> [1] | Υ | | | | |
| Derived PK Parameters | <b>Y</b> [3] | Υ | <b>Y</b> [3] | Υ | | Υ | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Tmax and tlag are not log transformed.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Mean (+SD) and Median plots will be generated.
- 3. Individual and Box Plot of DTG and RPV PK Parameters by Treatment

### 8.1.2. Endpoint / Variables

#### 8.1.2.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.4.3 Reporting Standards for Pharmacokinetic)

#### 8.1.2.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin 6.3 or higher. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve (AUC) from time 0 (predose) to time of the last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-24) | Area under the concentration-time curve (AUC) over time 0 (predose) to 24 hours |

| AUC(0-72) Area un after do: increme AUC(0-∞) Area un | se administration, to be calculated using the linear trapezoidal rule for each ental trapezoid and the log trapezoidal rule for each decremental trapezoid. der the concentration-time curve (AUC) over time 0 (predose) to 72 hours se administration, to be calculated using the linear trapezoidal rule for each ental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
|---|---|
| after do:<br>increme<br>AUC(0-∞) Area un | se administration, to be calculated using the linear trapezoidal rule for each ental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| \ / | |
| | der the concentration-time curve from time 0 (predose) extrapolated to ime, calculated as: |
| | $AUC(0-\infty) = AUC(0-t) + Ct / \lambda z$ |
| where C | It is the last observed quantifiable concentration. |
| %AUCex The per as: | centage of AUC(0-∞) obtained by extrapolation (%AUCex) will be calculated |
| [AUC(0- | ·∞) – AUC(0-t)] / AUC(0-∞) x 100 |
| Cmax Maximu data. | m observed concentration, determined directly from the concentration-time |
| Ct The last | observed quantifiable concentration |
| C24 The obs | served concentration at 24 hours after dose administration |
| t time of I | ast quantifiable concentration |
| Tmax Time to | first occurrence of Cmax |
| Tlast Time of | last quantifiable concentration |
| tlag Lag time | e before observation of drug concentrations in sampled matrix |
| t½ Termina | al phase half-life will be calculated as: |
| t½ = In2 | / λz |
| λz Termina | al-phase rate constant |
| CL/F The app | parent oral clearance |
| Vz/F The app | parent volume of distribution during the terminal phase |

#### NOTES:

• Additional parameters may be included as required.

# 8.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

# 8.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.2 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

For each of the Plasma DTG and RPV parameters  $AUC_{(0-\infty)}$ ,  $AUC_{(0-t)}$ ,  $C_{max}$ ,  $t_{lag}$ ,  $t_{max}$ ,  $t_{lag}$ ,  $\lambda z$ , % $AUC_{ex}$ ,  $AUC_{(0-24)}$ ,  $AUC_{(0-72)}$ , CL/F and Vz/F,  $C_t$ , and  $C_{24}$ , the following summary statistics will be calculated and tabulated by treatment (dose):

- Untransformed Data: N, n, arithmetic mean, %CV, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, and maximum.
- Loge-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of loge-transformed data and %CVb

For %AUCex, Tmax, tlag,  $\lambda z$ , t and Vz/F, the summary statistics specified for untransformed data above will be generated.

PK data will be listed and may be presented in graphical format and will be summarized descriptively. All PK data will be stored in the Archives, GlaxoSmithKline R& D. Statistical analyses of the PK parameter data will be the responsibility of Clinical Statistics, GlaxoSmithKline or their designee.

# 9. REFERENCES

GlaxoSmithKline Document Number 2018N392977\_00: A Phase I, Open-label, Single-dose Study to Investigate the Pharmacokinetics, Safety and Tolerability of Dolutegravir + Rilpivirine (JULUCA<sup>TM</sup>) 50 mg/25 mg tablets in healthy participants of Japanese descent. Effective Date: 04-APR-2019

# 10. APPENDICES

# 10.1. Appendix 1: Protocol Deviation Management and Definitions

Please refer to the Protocol Deviation Management Plan (PDMP).

# 10.1.1. Exclusions from PK Population

A subject meeting any of the following criteria will be excluded from the PK population:

| Number | Exclusion Description |
|--------|-------------------------------------------------------------|
| 01 | A subject with emesis occurring within 10 hours of the dose |

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

| | | Study Intervention Period | | | | | | | | | | Foll | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Da<br>y -<br>1 | Day | | | | | | | | | | ow- | |
| | | 1 | | | 2 | 3 | 4 | 6 | 8 | 10 | 12 | Up<br>(12 - | |
| Procedure | | Pr<br>e<br>D<br>os<br>e | 0<br>h<br>r | Post<br>Dose | 2<br>4<br>h<br>r | 4<br>8<br>hr | ~<br>7<br>2<br>hr | ~<br>1<br>2<br>0<br>hr | ~1<br>68<br>hr | ~2<br>16<br>hr | ~2<br>64<br>hr | 17 days post last dos e) 2,3 | Notes |
| Admission to Unit | Χ | | | | | | | | | | | | |
| Discharge | | | | | | Χ | | | | | | | |
| Outpatient Visit | | | | | | | Х | Χ | Χ | Χ | Χ | X | |
| Brief Physical<br>Exam <sup>1</sup> | Х | | | | | | | | | | | | |
| Pregnancy test (urine or serum) | Х | | | | | | | | | | | Х | |
| Urine/Drug/Alcohol/<br>Cotinine | Х | | | | | | | | | | | | Illicit Drug/Alcohol/Cotini ne performed at the standard practice of the site. |
| 12-Lead ECG | Χ | | | | | | | | | | | | Single ECGs will be collected |
| Vital Signs (VS) measurements | Х | Х | | | | | | | | | | Х | Single VS<br>measurements will<br>be performed at all<br>time points. |
| Safety lab<br>assessments<br>(Hematology,Chem<br>istry) | Х | | | | | Х | | | | | | | Glucose fasting is required approximately 10 hours prior to dosing on Day -1 and at least 6 hours at Day 3 post dose. |
| DTG/RPV FDC<br>Dosing | | | x | | | | | | | | | | Subjects will fast for ~10 hours and receive the dose ~30 minutes (± 5 minutes) after the start of a standardized moderate fat breakfast |

| | | Study Intervention Period Day | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Da<br>y -<br>1 | 1 | | | 2 | 3 | 4 | 6 | 8 | 10 | 12 | Up<br>(12 - | |
| Procedure | | Pr<br>e<br>D<br>os<br>e | 0<br>h<br>r | Post<br>Dose | 2<br>4<br>h<br>r | 4<br>8<br>hr | ~<br>7<br>2<br>hr | ~<br>1<br>2<br>0<br>hr | ~1<br>68<br>hr | ~2<br>16<br>hr | ~2<br>64<br>hr | days post last dos e) 2,3 | Notes |
| Pharmacokinetic<br>Sampling | | X | | Collected at 0.5,<br>1, 1.5, 2, 2.5, 3,<br>3.5, 4, 5, 6, 7, 8,<br>9, 12, 16, 24,<br>and 48 hours<br>post-dose | | | x | X | x | x | X | | Subjects should be scheduled to provide PK samples in the morning on Days 4, 6, 8, 10, and 12; Days 8, 10, and 12 are for RPV sampling only. The 4-hour post-dose sample must be drawn prior to the subjects' first post-dose meal |
| SAE Review | Χ | <b>-</b> | ←======X======X | | | | | | Χ | | | | |
| AE Review | | <del>(</del> = | ←======X======= | | | | | | Χ | | | | |
| Concomitant medication review | Χ | <del>(</del> = | === | | | | | | <b>⟨===</b> = | ==== | === | Χ | |

# 10.3. Appendix 3: Study Phases

# 10.3.1. Study Phases

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date ≤ Date ≤ Study Treatment Stop Date [+ 3 days] |
| Post-Treatment | Date > Study Treatment Stop Date [+ 3 days] |

### 1. NOTES:

If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

# 10.3.2. Study Phases for AE Data

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Event Start Date < Initial Study Treatment Date |
| On-Treatment | If event onset date is on or after the initial treatment date & on or before the final treatment date with 3 days lag time. Initial Study Treatment Date ≤ Event Start Date ≤ Final Study Treatment Date + 3 days |
| Post-Treatment | If event onset date is after the final treatment date with 3 days lag time. Event Start Date > Final Study Treatment Date + 3 days |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Date > Event Onset Date = Event Onset Date – Treatment Date If Treatment Date ≤ Event Onset Date = Event Onset Date – Treatment Date+1 Missing otherwise. |
| Duration (Days) | Event Resolution Date – Event Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing. |

### NOTES:

• If the initial and final study treatment dates are missing then the event will be considered to be On-Treatment.

# 10.4. Appendix 4: Data Display Standards & Handling Conventions

# 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | Reporting Area |
| HARP Server | : US1SALX00259-HARP PROD-US |
| HARP Compound | : GSK3365791 |
| Analysis Datasets | |
| Analysis datasets will be created according to Clinical Data Interchange Standards Consortium (CDISC) standards (SDTM IG Version 3.2 & Analysis Data Model (ADaM) Implementation Guide (ADaM IG) Version 1.0 or higher dataset standards) | |
| Generation of RTF Files | |
| RTF files will be generated for summary displays. | |

### 10.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and/or figures.
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 10.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [Insert document name]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Parameter Derivation | |
| PK Parameter to be<br>Derived by CPMS | The following PK parameters will be derived by the CPMS: Plasma DTG and RPV $AUC_{(0-\infty)}$ , $AUC_{(0-t)}$ , $C_{max}$ , $t_{lag}$ , $t_{max}$ , $t$ , $t_{1/2}$ , $\lambda z$ , % $AUC_{ex}$ , $AUC_{(0-24)}$ , $AUC_{(0-72)}$ , $CL/F$ and $Vz/F$ , $C_t$ , and $C_{24}$ |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Refer to [Standards for Handling NQ Impacted PK Parameters]. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. |

# 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

# 10.5.2. Study Population

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Only the year of birth will be collected. The date and month will be imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

### 10.5.3. Safety

#### **Adverse Events**

#### **AE'S of Special Interest**

No analysis for AEs of Special Interest will be performed.

### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

If ECGs are manually read, the RR value preceding the measurement QT interval should be a

### **ECG Parameters**

collected value THEN do not derive.

• Machine read values of RR should not be replaced with derived values.

### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as if he/she has completed all phases of the study including the last visit or the last scheduled procedure as shown in the Schedule of Activities.</li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start</li> </ul> </li> </ul> |
| | date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events. |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

# 10.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|-------------|-----------------------------------------|
| Concomitant | · |
| Medications | imputed using the following convention: |

| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
|---|---|
| AEs | <ul> <li>Any partial dates for AEs will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.7. Appendix 7: Values of Potential Clinical Importance

# 10.7.1. Laboratory Values

# 10.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | • | | |
| Absolute QTc Interval | msec | | > 450[1] |
| Absolute PR Interval | msec | < 110[1] | > 220[1] |
| Absolute QRS Interval | msec | < 75[1] | > 110 <sup>[1]</sup> |

### NOTES:

# 10.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

<sup>1.</sup> Represent standard ECG values of PCI for HIV studies.

# 10.8. Appendix 8: Abbreviations & Trade Marks

# 10.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| ADaM IG | Analysis Data Model Implementation Guide |
| AE | Adverse Event |
| AUC | Area under the concentration-time curve |
| AUC(0-t) | Area under the concentration-time curve from time 0 (predose) to time |
| | of the last quantifiable concentration |
| AUC(0-24) | Area under the concentration-time curve over time 0 (predose) to 24 |
| , , , | hours after dose administration |
| AUC(0-72) | Area under the concentration-time curve over time 0 (predose) to 72 |
| | hours after dose administration |
| $AUC(0-\infty)$ | Area under the concentration-time curve from time 0 (predose) |
| | extrapolated to infinite time |
| %AUCex | The percentage of AUC( $0-\infty$ ) obtained by extrapolation |
| BMI | Body Mass Index |
| C24 | The observed concentration at 24 hours after dose administration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CL/F | The apparent oral clearance |
| Cmax | Maximum observed concentration |
| CI | Confidence Interval |
| Ct | The last observed quantifiable concentration |
| CTMS | Clinical Trial Management System |
| CV | Coefficient of variation |
| $CV_b$ | Coefficient of variation (Between) |
| DAIDS | Division of Acquired Immune Deficiency Syndrome |
| DTG | Dolutegravir |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| GSK | GlaxoSmithKline |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| kg | Kilograms |
| m | Meters |
| mg | Milligrams |
| msec | Milliseconds |
| PK | Pharmacokinetic |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| R&D | Research and Development |
| RAP | Reporting & Analysis Plan |
| RPV | Rilpivirine |
| SAC | Statistical Analysis Complete |

| Abbreviation | Description |
|---|---|
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| t | Time of last quantifiable concentration |
| TFL | Tables, Figures & Listings |
| t½ | Terminal phase half-life |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| Tlast | Time of last quantifiable concentration |
| Tmax | Time to first occurrence of Cmax |
| Vz/F | The apparent volume of distribution during the terminal phase |
| $\lambda z$ | terminal phase rate constant |

# 10.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| JULUCA |
| TIVICAY |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| DAIDS |
| EDURANT |
| SAS |
| WinNonlin |

# 10.9. Appendix 9: List of Data Displays

# 10.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.7 | N/A |
| Safety | 3.1 to 3.13 | N/A |
| Pharmacokinetic | 4.1 to 4.6 | 4.1 to 4.10 |
| Section | List | ings |
| ICH Listings | 1 to 29 | |
| Other Listings | 30 to | o 33 |

# 10.9.2. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [1] | Final Statistical Analysis Complete |

### NOTES:

<sup>1.</sup> Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 10.9.3. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | Safety | ES1 | Summary of Participant Disposition for the Participant Conclusion Record | | SAC [1] |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | | SAC [1] |
| 1.3. | Screened | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| 1.4. | Safety | DM1 | Summary of Demographic Characteristics | | SAC [1] |
| 1.5. | Enrolled | DM11 | Summary of Age Ranges | | SAC [1] |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |
| Prior a | Prior and Concomitant Medications | | | | |
| 1.7. | Safety | MH1 /<br>MH4 | Summary of Current Medical Conditions | | SAC [1] |

# 10.9.4. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | • | • |
| 3.1. | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC [1] |
| 3.2. | Safety | AE1 | Summary All Drug-Related Adverse Events | | SAC [1] |
| 3.3. | Safety | AE5a | Summary of Adverse Events by Maximum Grade by System Organ Class and Preferred Term | | SAC [1] |
| Labora | tory: Chemistry | у | | | |
| 3.4. | Safety | LB1 | Summary of Chemistry Values | | SAC [1] |
| 3.5. | Safety | LB1 | Summary of Chemistry Changes from Baseline | Add Footnote - Note: Baseline is defined as Day -1 | SAC [1] |
| 3.6. | Safety | LB16 | Summary of Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC [1] |
| Labora | tory: Hematolo | gy | | | |
| 3.7. | Safety | LB1 | Summary of Hematology Values | | SAC [1] |
| 3.8. | Safety | LB1 | Summary of Hematology Changes from Baseline | Add Footnote - Note: Baseline is defined as Day -1 | SAC [1] |
| 3.9. | Safety | LB16 | Summary of Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC [1] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborat | ory: Urinalysis | | | | |
| 3.10. | Safety | LB1 | Summary of Urinalysis Dipstick Results | | SAC [1] |
| Laborat | ory: ECG | | | | |
| 3.11. | Safety | EG1 | Summary of ECG Findings | | SAC [1] |
| Vital Sig | Vital Signs | | | | |
| 3.12. | Safety | VS1 | Summary of Vital Signs | | SAC [1] |
| 3.13. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | Add Footnote - Note: Baseline is defined as Day 1 (Predose) | SAC [1] |

# 10.9.5. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | centration Dat | a | | | |
| 4.1. | PK | PKCT1 | Summary of DTG Plasma Pharmacokinetic Concentration-Time Data by Treatment | | SAC [1] |
| 4.2. | PK | PKCT1 | Summary of RPV Plasma Pharmacokinetic Concentration-Time Data by Treatment | | SAC [1] |
| PK Der | ived Parameter | 'S | | | |
| 4.3. | PK | PKPT1 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (Non-Transformed) by Treatment | Parameters with units | SAC [1] |
| 4.4. | PK | PKPT3 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (Loge-transformed) by Treatment | Parameters with units | SAC [1] |
| 4.5. | PK | PKPT1 | Summary of Derived RPV Plasma Pharmacokinetic Parameters (Non-Transformed) by Treatment | Parameters with units | SAC [1] |
| 4.6. | PK | PKPT3 | Summary of Derived RPV Plasma Pharmacokinetic Parameters (Loge-transformed) by Treatment | Parameters with units | SAC [1] |

# 10.9.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentrati | ion Plots | | | • |
| 4.1. | PK | PKCF1 | Individual participant DTG Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant | SAC [1] |
| 4.2. | PK | PKCF1 | Individual participant RPV Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant | SAC [1] |
| 4.3. | PK | PKCF6 | Individual participant DTG Plasma Concentration-Time Plots by treatment (Linear and Semi-Logarithmic) | Only 1 page as one Treatment group | SAC [1] |
| 4.4. | PK | PKCF6 | Individual participant RPV Plasma Concentration-Time Plots by treatment (Linear and Semi-Logarithmic) | Only 1 page as one Treatment group | SAC [1] |
| Mean / | Median Conce | ntration Plots | | | • |
| 4.5. | PK | PKCF2 | Arithmetic Mean DTG Plasma Concentration-time Plot (Linear and Semi-log) | Use nominal times in X Axis, | SAC [1] |
| 4.6. | PK | PKCF2 | Arithmetic Mean RPV Plasma Concentration-time Plot (Linear and Semi-log) | Use nominal times in X Axis, | SAC [1] |
| 4.7. | PK | PKCF3 | Median DTG Plasma Concentration-time Plot (Linear and Semilog) | Use nominal times in X Axis, | SAC [1] |
| 4.8. | PK | PKCF3 | Median RPV Plasma Concentration-time Plot (Linear and Semilog) | Use nominal times in X Axis, | SAC [1] |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Der | ived Parameter | rs | | | |
| 4.9 | PK | Figure 3.19<br>201674 | Individual and Box Plot of DTG PK Parameters by Treatment | AUC(0-∞), AUC(0-24), AUC(0-72),<br>AUC(0-t), %AUCex, CL/F, C24,<br>Cmax, t½, tlag, tlast,<br>tmax, Vz/F | SAC [1] |
| 4.10 | PK | Figure 3.19<br>201674 | Individual and Box Plot of RPV PK Parameters by Treatment | AUC(0-∞), AUC(0-24), AUC(0-72),<br>AUC(0-t), %AUCex, CL/F, C24,<br>Cmax, t½, tlag, tlast,<br>tmax, Vz/F | SAC [1] |

# 10.9.7. ICH Listings

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Subject Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC [1] |
| 2. | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3. | Safety | TA1 / CP_RD1x | Listing of Planned and Actual Treatments | | SAC [1] |
| Protoc | ol Deviations | | | | |
| 4. | Safety | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 5. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| Popula | tions Analysed | | | | |
| 6. | Screening | SP3 | Listing of Participants Excluded from Any Population | | SAC [1] |
| Demog | raphy | | | | |
| 7. | Safety | DM4 | Listing of Demographic Characteristics | | SAC [1] |
| 8. | Safety | DM10 | Listing of Race | | SAC [1] |
| Prior a | nd Concomitan | t Medications | | | |
| 9. | Safety | CP_CM4 | Listing of Concomitant Medications | | SAC [1] |
| Exposure | | | | | |
| 10. | Safety | EX34 | Listing of Exposure Data | | SAC [1] |
| Advers | Adverse Events | | | | |
| 11. | Safety | CP_AE9 | Listing of All Adverse Events | | SAC [1] |
| 12. | Safety | CP_AE9 | Listing of Drug Related Adverse Events | | SAC [1] |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 13. | Safety | AE8 | Listing of Non-Serious Adverse Events | | SAC [1] |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [1] |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC [1] |
| Serious | s and Other Sig | nificant Adverse | Events | | |
| 16. | Safety | CP_AE9 | Listing of Adverse Events Leading to Withdrawal from study | | SAC [1] |
| 17. | Safety | CP_AE9a | Listing of Serious Adverse Events | | SAC [1] |
| All Lab | oratory | | | | |
| 18. | Safety | LB6 | Listing of Clinical Chemistry Toxicities of all Lab Abnormalities | | SAC [1] |
| 19. | Safety | LB6 | Listing of All Clinical Chemistry Data for Participants with Lab Abnormalities | | SAC [1] |
| 20. | Safety | LB6 | Listing of Hematology Toxicities of all Lab Abnormalities | | SAC [1] |
| 21. | Safety | LB6 | Listing of All Hematology Data for Participants with Lab Abnormalities | | SAC [1] |
| 22. | Safety | LB6 | Listing of Urinalysis Data for Subjects with Positive Dipstick or Microscopic Results | | SAC [1] |
| ECG | | | | | |
| 23. | Safety | EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | | SAC [1] |
| 24. | | | Listing of ECG Values of Potential Clinical Importance | | |
| 25. | Safety | EG6 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | | SAC [1] |
| 26. | Safety | EG6 | Listing of Abnormal ECG Findings | | SAC [1] |
| Vital Si | gns | | | | |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 27. | Safety | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | | SAC [1] |
| 28. | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance | | |
| Liver Events | | | | | |
| 29. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC[1] |

# 10.9.8. Non-ICH Listings

| Non-ICI | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | PK | | | | |
| 30. | PK | PKCL1X | Listing of DTG Plasma Pharmacokinetic Concentration-Time Data | | SAC [1] |
| 31. | PK | PKCL1X | Listing of RPV Plasma Pharmacokinetic Concentration-Time Data | | SAC [1] |
| 32. | PK | PKPL1X | Listing of Derived DTG Plasma PK Parameters | | SAC [1] |
| 33. | PK | PKPL1X | Listing of Derived RPV Plasma PK Parameters | | SAC [1] |